CLINICAL TRIAL: NCT05996393
Title: Ciclosporin + Antithymocyte Immunoglobulin + Avatrombpag Versus Ciclosporin + Avatrombpag for the Treatment of Severe Aplastic Anemia in the Elderly
Brief Title: CsA+ATG+AVA vs. CsA+AVA for the Treatment of Newly-diagnosed SAA in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVA-3
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclosporine; avatrombopag; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CsA+ATG+AVA (Experimental): Ciclosporine: 3-5 mg/kg/d orally, with ciclosporine trough concentrations maintained at 100-200 ng/ml for 3 months to achieve maximum efficacy and then tapered; Anti-human thymocyte: rabbit anti-human thymocyte globulin (r-ATG 3mg/kg/d) was administered intravenously for 5 days; Avatrombopag:60 mg/d orally, for a total of 24 weeks. Adjust the dose according to the platelet counts of patients.
  Interventions: Drug: Ciclosporin; Drug: Avatrombopag; Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit
- CsA+AVA (Experimental): Ciclosporine: 3-5 mg/kg/d orally, with ciclosporine trough concentrations maintained at 100-200 ng/ml for 3 months to achieve maximum efficacy and then tapered; Avatrombopag:60 mg/d orally, for a total of 24 weeks. Adjust the dose according to the platelet counts of patients.
  Interventions: Drug: Ciclosporin; Drug: Avatrombopag

INTERVENTIONS:
Drug: Ciclosporin — 3-5 mg/kg/d orally, trough concentrations: 100-200 ng/ml
Drug: Avatrombopag — 60 mg/d orally, 24 weeks
Drug: Anti-Human Thymocyte Immunoglobulin, Rabbit — rabbit anti-human thymocyte immunoglobulin (r-ATG 3mg/kg/d), intravenously, 5 days;
  Arms: CsA+ATG+AVA

SUMMARY:
This is a multicenter, prospective, randonmized study. Our previous retrospective study showed that for SAA patients who were intolerant to ATG, CsA+ eltrombopag (EPAG) had similar efficacy to CsA+ATG+EPAG. Since the action mechanism of AVA and EPAG is not exactly the same, and the metabolic level of the elderly is not the same as that of younger patients, it is unknown whether there are predictive factors of efficacy in the treatment of AVA. We wondered whether CsA+AVA could achieve an efficacy similar to CsA+ATG+AVA in the Elderly. Meanwhile, to explore the predictive factors of efficacy, to find out a safe and effective treatment strategy for the Elderly.

DETAILED DESCRIPTION:
Aplastic anemia (AA) can be divided into severe AA (SAA) and non-severe AA (NSAA), according to the severity of the disease. For SAA patients with o condition of hematopoietic stem cell transplantation, guideline recommended ciclosporin A (CsA) + anti-thymocyte immunoglobulin (ATG) + thrombopoietin receptor agonists (TPO-RA) as the first-line therapy. Our previous retrospective study showed that for SAA patients who were intolerant to ATG, CsA+ eltrombopag (EPAG) had similar efficacy to CsA+ATG+EPAG. However, the adverse effects such as hepatotoxicity and gasrointestinal disorder limit its application in elderly SAA.Compared with EPAG, AVA has no hepatotoxicity and less other adverse effects, but there was few studies for AA. Our previous study demonstrated that AVA was effective in 55% of refractory AA. Since the action mechanism of AVA and EPAG is not exactly the same, and the metabolic level of the elderly is not the same as that of younger patients, it is unknown whether there are predictive factors of efficacy in the treatment of AVA. Thus, we wondered whether CsA+AVA could achieve an efficacy similar to CsA+ATG+AVA in the Elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed severe aplastic anemia, aged greater than 60 years.
2. Patients met the diagnostic criteria of severe aplastic anemia (SAA).
3. Complete all screening assessments as outlined in the test protocol.
4. Without or with no more than 1 month treatment of ciclosporine, tacrolimus, glucocortocoid, or TPO-RAs.
5. Agree to sign the informed consent form.

Exclusion Criteria:

1. Known diagnosis of congenital hematopoietic failure disorders (e.g. Fanconi anemia) and other causes of cytopenia.
2. Patients with uncontrolled bleeding and/or infection despite standard treatment.
3. Patients with previous history of hematopoietic stem cell transplantation.
4. Patients with previous history of thrombosis in 1 year.
5. Patients with concurrent malignancy.
6. Those who are considered unsuitable for enrollment by the investigator.
7. Abnormal renal function: creatinine > 1.2 normal upper limit, albumin < 0.9 normal lower limit, or CLcr < 30 ml/min.
8. Abnormal liver function: transaminase > 2.5 normal upper limit, or tota bilirubin > 2.5 normal upper limit.
9. Patients with severe heart, liver or renal disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 6 month
  Proportion of patient who achieved partial response or complete response

SECONDARY OUTCOMES:
Complete response rate | 6 month
  Proportion of patient who achieved complete response (HGB>100g/L, PLT>100×109/L, ANC>1.0×109/L)
Relapse rate | 12 month
  Proportion of patient who relapse
Adverse event rate | 3, 6, 12 month
  Proportion of patient who adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Tang Z, Huang Y, Hu Q, Wang S, Ji J, Du Y, Yang C, Chen M, Hu S, Han B. Sirolimus versus cyclosporine A in patients with primary acquired pure red cell aplasia: a prospective cohort study. Blood Cancer J. 2023 May 10;13(1):74. doi: 10.1038/s41408-023-00845-3. No abstract available. PMID 37160872
- [Background] Chi Y, Hu Q, Yang C, Chen M, Han B. Avatrombopag is effective in patients with chemoradiotherapy-induced aplastic anemia: a single-center, retrospective study. Exp Hematol. 2023 Jan;117:62-68. doi: 10.1016/j.exphem.2022.11.002. Epub 2022 Nov 16. PMID 36400314
- [Background] Wan Z, Chen M, Han B. Avatrombopag, a promising novel thrombopoietin receptor agonist for refractory/relapsed/intolerant non-severe aplastic anemia: a phase 2 single-arm clinical trial. Ann Med. 2023 Dec;55(1):2224044. doi: 10.1080/07853890.2023.2224044. PMID 37318085
- [Background] Chen F, Hu S, Ruan J, Chen M, Han B. Mutational landscape and its clinical significance in paroxysmal nocturnal hemoglobinuria. Blood Cancer J. 2021 Mar 16;11(3):58. doi: 10.1038/s41408-021-00451-1. No abstract available. PMID 33727526
- [Background] Chen M, Liu Q, Gao Y, Suo X, Ding X, Wang L, Li L, Shao Y, Gao D, Sun W, Tan Y, Wang W, Ye F, Han B. Cyclosporine plus eltrombopag in the treatment of aplastic anemia with or without antithymocyte immunoglobulin: A multicenter real-world retrospective study. Eur J Haematol. 2023 Sep;111(3):407-413. doi: 10.1111/ejh.14021. Epub 2023 Jun 4. PMID 37271577